CLINICAL TRIAL: NCT04527042
Title: Effectiveness and Safety of Rivaroxaban Used in Clinical Practice of Extended Anticoagulation for Pulmonary Embolism Patients in China, XAPEC-EXT
Brief Title: Effectiveness and Safety of Rivaroxaban Used in Extended Anticoagulation for Pulmonary Embolism Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Deputy Director of the Second Department of Respiratory and Critical Care Medicine, China-Japan Friendship Hospital
Other Study IDs: CJFH-2020-PE-ZZG
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Embolism
Keywords: Clinical Practice of Extended Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban — It is determined by the clinician's routine clinical prescription.
  Other Names: XARELTO

SUMMARY:
Domestic and international guidelines for the management of pulmonary embolism have suggested that the standard duration of anticoagulation should cover at least 3 months.Whether extended anticogulation therapy shoud balance the efficacy and safety of the therapy.Nevertheless, the concerning about bleeding may affect the decision on the extended anticoagulation for pulmonary embolism patients who may benefit from continuing anticoagulation. Rivaroxaban is an oral direct factor Xa inhibitor, it does not require routine laboratory monitoring and has no food interactions and only a few drug interactions compared to standard of care with the recommendation for the treatment of pulmonary embolism by several guidelines.Our study aims to acquire the data of effectiveness and safety of rivaroxaban used in clinical practice of extended anticoagulation for pulmonary embolism patients in China through this perspective observational study.

DETAILED DESCRIPTION:
This is a perspective, multicenter, single-arm, non-interventional, and observational study. The primary objective is to evaluate the effectiveness and safety of rivaroxaban used in extended treatment of pulmonary embolism in a real-world.The secondary objective aims to analyze the drug usage pattern of rivaroxaban, patient satisfaction and medical resource utilization used in extended treatment of pulmonary embolism in a real-world.496 subjects will be enrolled in this study. The primary outcome of this study is net clinical benefit.

All patients with rivaroxaban should be followed up to 12 months, or about 30 days after the end of rivaroxaban treatment if discontinued before the completion of 12 months. Follow up visits occur at initial visit, 3, 6, 9, 12 months after the initial visit, where such data have been collected as part of routine clinical practice, by phone and or face to face interview.

During each follow up visit, the date of visit, physical examination, ACTS and, as applicable, changes in the concomitant medication, changes in concomitant disease,changes in pulmonary embolism and/or treatment regimen, new diagnosis of venous thromboembolism, medical resources utilization, and adverse events will be obtained and recorded.

Starting with the first application of rivaroxaban after enrollment into the study or follow-up period, all AEs would be documented. For each AE, the investigator must assess and document the seriousness, duration, relationship to product, action taken and outcome of the event.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 years or above
2. Objectively confirmed diagnosis of symptomatic or asymptomatic pulmonary embolism
3. Already received 6 to 12 months anticoagulant
4. Indication for extend anticoagulant for at least 3 months with rivaroxaban( as assessed by the investigator)5)Written informed consent

Exclusion Criteria:

1. Patients with another indication for anticoagulation other than venous thromboembolism.
2. Patients with contraindications listed in rivaroxaban label in china.
3. Patients who participated in another study within 30 days
4. Life expectation less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary Embolism patients
Sampling Method: Non-Probability Sample
Enrollment: 496 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-11-29 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Net clinical benefit | 12 months
  Net clinical benefit(the composite of major bleeding and symptomatic recurrent venous thromboembolism)

SECONDARY OUTCOMES:
The symptomatic recurrent venous thromboembolism | 12 months
  The symptomatic recurrent venous thromboembolism, is the composite of recurrent deep vein thrombosis or fatal or non-fatal pulmonary embolism.
Major bleeding | 12 months
  Major bleeding was defined as overt bleeding and: associated with a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or occurring in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or contributing to death.
Clinical related non-major bleeding events | 12 months
  Clinical related non-major bleeding events: other dominant bleeding, which does not conform to the criteria for major bleeding, but requires medical intervention; an unscheduled contact with a doctor either through telephone or through face-to-face interview, temporary stop of the treatment, or other discomforts, such as pain.
Mortality | 12 months
  All-cause mortality
The satisfaction with anticoagulant treatment | 12 months
  The Anti-Clot Treatment Scale (ACTS) is a 17-item patient-reported instrument of satisfaction with anticoagulant treatment.
Length of stay in hospital | 12 months
  Medical resources utilization
The number of outpatient visits | 12 months
  Medical resources utilization
Medical costs due to bleeding or embolism | 12 months
  Medical resources utilization
Drug use patterns | 12 months
  Drug use patterns (including dosage of rivaroxaban, course of treatment, reasons for withdrawal/interruption/dressing change, combined medication)
Adverse events | 12 months
  Adverse events (AEs) and serious adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, Ph.D, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No